CLINICAL TRIAL: NCT05037955
Title: Follow-up Assessment of Rhinitis - Quality of Life in Allergic Patients Treated With Intralymphatic Immunotherapy (ILIT)
Brief Title: ILIT: Follow-up of Rhinitis Quality of Life
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Pal Johansen, Professor, PhD, University of Zurich
Other Study IDs: 2020-02369
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Allergic Rhinitis Due to Grass Pollen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ILIT from trial NCT00470457: Patients who received ILIT in the original trial in 2005
- SCIT from trial NCT00470457: Patients who received SCIT in the original trial in 2005
- SCIT outpatient control: Patients who visited the allergy unit at the University Hospital Zurich and completed SCIT in the last 5 years

SUMMARY:
Re-evaluation of patients treated with intralymphatic immunotherapy (ILIT) in terms of quality of life and therapeutic efficacy and comparison with subcutaneous immunotherapy (SCIT) 15 years post immunotherapy

DETAILED DESCRIPTION:
In Switzerland, around 20% of the population suffers from hay fever. The allergy usually begins in childhood and can worsen or improve as the child grows. The quality of life of those affected suffers greatly. Since the allergens are seasonally found in the air, patients cannot really avoid the source of the allergy. On the one hand, allergic rhinitis can be treated pharmacologically. On the other hand allergen-specific immunotherapy (AIT) (=desensitization), can be considered. AIT can greatly reduce the symptoms and restore the patient's quality of life. It is the only treatment method that can offer long-term therapeutic success without the need for regular medication.

Subcutaneous immunotherapy (SCIT) is the traditional method in which the allergen is administered subcutaneously over a period of three to four years with alternating treatment intervals. The chances of success are good, but the drop-out rate is comparatively high due to the long treatment period (at least 3 and up to 5 years). In contrast, intralymphatic immunotherapy (ILIT) requires only three sessions over a period of three to four months. The allergen is administered by ultrasound directly into a lymph node. The results are equally good (compared to SCIT), but the treatment time is much shorter.

In the following project, the quality of life of the people who participated in the first ever ILIT study (ClinicalTrials.gov Identifier: NCT00470457) will be evaluated. The aim is to have a meaningful result on the duration of the therapeutic effect, as judged by the patients themselves.

To develop a meaningful result, a questionnaire was designed for patients to fill out at baseline (prior to pollen season). This shold allow assessmen of how each individual's quality of life has evolved since treatment. The study subjects will also receive a standardised (European) questionnaire. This questionnaire refers to the quality of life and symptoms of the last seven days and is filled out at baseline (prior to season) and in season (Mai-June). The data will be analysed and presented to the scientific and clinical audience as soon as possible.

ELIGIBILITY:
Inclusion Criteria:

* Receiving ILIT or SCIT treatment at the USZ.
* Indication: hay fever (type I sensitisation to grass pollen)
* Adult male and female patients
* Written/digital informed consent of the participating person
* Complete return of both questionnaires

Exclusion Criteria:

* Discontinuation of immunotherapy
* Incomplete data set
* Pathological barrier (e.g. dementia)
* Language barrier (not understanding the German language)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male and female patients with past or current hay fever due to grass pollen sensitisation. The patients received immunotherapy (SCIT or ILIT) in the NCT00470457 trials from 2005. A control group of patients received and completed SCIT as standard treatment of their hay fever at the Allergy Unit of the University Hospital Zurich during the last five years.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Rhinoconjunctivitis quality of life | February 2021 through June 2021
  The standardised scoring of the outcomes "activities", "sleep", "non-nose/eye symptoms", "practical problems", "nasal symptoms", "eye symptoms", and "emotional" are entered in the form names "Rhinoconjunctivitis quality of life questionnaire with standardised activities (RQLQ)". The scoring is from 0 ("not troubled" or "none of the time") to 6 ("extremely troubled" or "all of the time").

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No